CLINICAL TRIAL: NCT06551259
Title: Effect of Intraoperative Dextrometomidine on Complications of the Central Nervous System in Patients Undergoing Cardiac Surgery: a Randomized Controlled Trial
Brief Title: Effect of Dexmedetomidine on Central Nervous System Complications in Patients Undergoing Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PLAGH-DEX-RCT-01
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Randomized Controlled Trial; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group: dexmedetomidine (Experimental): Intravenous infusion of 0.6μg/kg load dose of dexmedetomidine within 10 minutes after intubation, followed by continuous infusion at a rate of 0.4 μg/kg/h until 30 minutes before the end of surgery
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): Provide equal volume of physiological saline
  Interventions: Drug: physiological saline

INTERVENTIONS:
Drug: Dexmedetomidine — Intravenous infusion of 0.6μg/kg load dose of dexmedetomidine within 10 minutes after intubation, followed by continuous infusion at a rate of 0.4 μg/kg/h until 30 minutes before the end of surgery
  Arms: Intervention group: dexmedetomidine
Drug: physiological saline — physiological saline
  Arms: Control group

SUMMARY:
With the continuous improvement of medical technology, more and more patients need to undergo surgery as a kind of treatment for their diseases. However, there are various pains that may occur in the perioperative period, risks associated with anesthesia, loss of body organs, surgical trauma, and postoperative procedures Factors such as the onset of the disease can cause the vast majority of patients to have varying degrees of emotional reactions such as worry, worry, nervousness, and fear. Emotional disorders such as depressed mood, disappointed crying, decreased mobility, and delayed thinking and cognitive function, that is, postoperative psychiatric symptoms.

Dexmedetomidine (DEX) is an alpha-2 adrenergic agonist that works by inhibiting norepinephrine. Releasing renaline, which reduces inflammation and thus plays a protective role in the central nervous system. Previous studies have shown that dexmedetomidine is lowering. DEX has the potential to prevent and treat patients undergoing cardiac surgery. The role of postoperative anxiety and depression needs to be further explored for evidence-based evidence. Based on the above research background, the hypothesis of this study is proposed. The intraoperative use of dexmedetomidine has a positive effect on alleviating postoperative anxiety and depression in patients undergoing postoperative cardiac surgery.

DETAILED DESCRIPTION:
1. Observing the effect of intraoperative use of dexmedetomidine on the incidence of postoperative anxiety and depression in patients undergoing cardiac surgery;
2. Observe the effects of intraoperative use of dexmedetomidine on postoperative delirium, quality of life, pain scores, and sleep quality in patients undergoing cardiac surgery;
3. To provide a feasible plan for preventing and treating postoperative anxiety and depression in patients undergoing cardiac surgery, improve the quality of patient prognosis, and reduce the burden on society.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 85 years old, regardless of gender
2. Patients who undergo cardiac surgery on a scheduled basis;
3. ASA level 1-4;
4. Obtain written informed consent form;

Exclusion Criteria:

1. Patients with MMSE scores less than 18 or dementia, intellectual disability, and inability to communicate (coma, severe dementia, hearing or language impairment);
2. Have a history of mental or neurological disorders (such as schizophrenia, epilepsy, Parkinson's disease, or severe myasthenia gravis);
3. Previous history of brain injury;
4. Severe liver dysfunction (Child pugh C-grade) or renal insufficiency (preoperative dialysis);
5. Severe bradycardia (heart rate below 50 beats per minute), pathological sinus syndrome, or atrioventricular block without a pacemaker;
6. Postoperative intensive care unit (ICU) duration exceeding 7 days or death;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative depression | Postoperative 7 days and 30 days
  Patient Health Questionnaire-9 (PHQ-9) scale assesses depressive symptoms

SECONDARY OUTCOMES:
The incidence of postoperative anxiety | Postoperative 7 days and 30 days
  Generalized Anxiety Disorder-7 (GAD-7) Scale to Assess Anxiety Symptoms
The incidence of postoperative delirium | Postoperative 7 days
  Patients in the 3-Minute Diagnostic Interview for CAM (3D-CAM) general ward are evaluated by 3D-CAM. Delirium consists of four main features: acute altered mental status or fluctuating levels of consciousness, difficulty concentrating, confusion, and altered levels of consciousness. If both the first and second features are present, and the third or fourth feature is present, the patient is diagnosed with postoperative delirium.
Postoperative Pain | Postoperative 7 days and 30 days
  NRS Pain Scoring Criteria (0-10): NRS is 0-10, with 0 indicating no pain and 10 indicating the worst pain. The total amount of analgesic drug consumption and the number of PCIA active compressions within 48 hours were recorded every day
Postoperative quality of life evaluation | Postoperative 30 days
  Five-dimensional health scale EQ-5D, the five-dimensional health scale consists of 5 dimensions: mobility, self-care, activities of daily living, pain or discomfort, anxiety or depression. Each dimension contains three levels: no difficulty, some difficulty, and extreme difficulty. Through the conversion of effect size, the respondents can make choices at the five dimensions and three levels in the questionnaire, and calculate the score of the five-dimensional health scale index.
Postoperative mortality rate | Postoperative 7 days and 30 days
  Follow-up by phone or mail for patient mortality.
Surgical related complications | Postoperative 7 days
  Surgery-related complications include cardiovascular, respiratory, pulmonary, digestive, urinary, neurological, infection, pain, and bleeding from the surgery.
Postoperative sleep quality | Postoperative 7 days and 30 days
  Postoperative sleep quality was measured using the Pittsburgh Sleep Quality Index scale.

CONTACTS AND LOCATIONS:
Overall Officials: WEIDONG MI, PhD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No